CLINICAL TRIAL: NCT03850184
Title: Translation of the "Exercise in Mental Illness Questionnaire (EMIQ) - Health Practicioners Version" From English to German
Brief Title: Translation of the "Exercise in Mental Illness Questionnaire (EMIQ)" to German
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Moritz Petzold, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: TEMIQG
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Physical Activity; Psychiatric Disorder
MeSH Terms: conditions — Motor Activity; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mental Health Professionals: Psychiatrists, Psychologists, Nurses working with patients with mental disorders
  Interventions: Diagnostic Test: The Exercise in Mental Illness Questionnaire (EMIQ)

INTERVENTIONS:
Diagnostic Test: The Exercise in Mental Illness Questionnaire (EMIQ) — Questionnaire assessing prescription behaviour, knowledge, barriers and behaviour of physical activity in mental health professionals

SUMMARY:
The "The Exercise in Mental Illness Questionnaire (EMIQ) - Health Practicioners Version" is a questionnaire designed to assess the prescription behaviour of physical activity as well as related knowledge, barriers and exercise behaviour of mental health professionals.

As a lot of research on prescription behaviour is done using unvalidated questionnaires we want to translate this validated questionnaire into German for further use in this research field.

DETAILED DESCRIPTION:
The "The Exercise in Mental Illness Questionnaire (EMIQ) - Health Practicioners Version" is a questionnaire designed to assess the prescription behaviour of physical activity as well as related knowledge, barriers and exercise behaviour of mental health professionals.

As a lot of research on prescription behaviour is done using unvalidated questionnaires we want to translate this validated questionnaire into German for further use in this research field. Therefore we plan to translate the questionnaire in accordance to established questionnaire translation guidelines.

Then we plan to validate the questionnaire in a sample of about 30 mental health professionals (psychiatrists, psychologists, nurses) currently working with patients with mental disorders. We plan to evaluate re-test-reliability using repeated measurement within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrist, Psychologist or Nurse
* Working with patients with mental disorders
* German mother language

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to evaluate the questionnaire in mental health professioals (psychiatrists, psychologists, nurses) currently working with patients with mental disorders
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
The Exercise in Mental Illness Questionnaire (EMIQ) | within 7 days
  Questionnaire assessing the following areas: knowledge, attitudes, beliefs and behavirous of physical activity in mental health professionals.
  Outcome in this validation study are the intra-class-correlations of the single items to assess re-test-reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz B Petzold, Dipl.-Psych., Principal Investigator — Charité University Medicine Berlin - Department of Psychiatry and Psychotherapy - CCM, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin - Departement of Psychiatry, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanton R, Happell B, Reaburn P. The development of a questionnaire to investigate the views of health professionals regarding exercise for the treatment of mental illness,. Mental Health and Physical Activity 7(3): 177-182, 2014.